CLINICAL TRIAL: NCT05830929
Title: Ovarian Tissue Cryopreservation and Subsequent Auto-Transplantation for Female Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023.096-T
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian tissue freezing and subsequent auto-transplantation after thawing (Experimental): Ovarian tissue freezing and subsequent auto-transplantation after thawing
  Interventions: Procedure: Ovarian tissue freezing and subsequent auto-transplantation after thawing

INTERVENTIONS:
Procedure: Ovarian tissue freezing and subsequent auto-transplantation after thawing — Removal of the ovarian tissue will be retrieved via laparoscopic surgery under general anesthesia. The ovarian cortical tissue obtained will be transferred on ice to the laboratory for cryopreservation. After medical treatment, if the patient would like to start a family but has experienced premature ovarian failure, she will have ovarian tissue auto-transplantation after thawing.

SUMMARY:
Ovarian Tissue Cryopreservation will be provided to cancer patients to allow them to have their fertility preserved.

DETAILED DESCRIPTION:
This project hopes to provide Ovarian Tissue Cryopreservation to patients who do not have adequate time for ovarian stimulation in oocyte or embryo freezing and in prepubertal girls where oocyte freezing is not possible. All the patients will have fertility preservation consultations with a fertility specialist in our unit to go through the details of ovarian Tissue Cryopreservation service and risks related to ovarian tissue cryopreservation procedures. After undergoing ovarian tissue collection via surgery, the collected ovarian tissue will be cryopreserved either by slow freezing or vitrification in our unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 0-35 years old and diagnosed with cancer e.g., leukaemia, myeloproliferative or myelodysplastic diseases, lymphoma, bone tumours, neurological neoplasms and sarcoma, Paediatric bone marrow transplant patients
* Patients with any illness or who will undergo any type of treatment that may cause irreversible damage to their fertility, such as extensive abdominal surgery, high toxicity medication and treatments;
* Patients suffering from hormone-sensitive malignancies who will undergo medical treatment, such as radiotherapy and chemotherapy that is liable to damage their ovaries and deter them from conception in the future.

Exclusion Criteria:

* Patients with no anticipated oncologic therapies
* Patients who are pregnant
* Children with one ovary
* Children deemed high risk for perioperative complications
* Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Ages: 1 Month to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2043-04-30 (Estimated); Study Completion 2043-12-30 (Estimated)

PRIMARY OUTCOMES:
Surgical complications | 15 years
  Surgical complications after ovarian tissue transplantation

SECONDARY OUTCOMES:
Pregnancy rate | 15 years
  Pregnancy rate after ovarian tissue transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pui Wah CHUNG, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No